CLINICAL TRIAL: NCT02517957
Title: Xia Shi Surgical Treatment for Eczema Multi-center Clinical Research
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14401970200
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Eczema
Keywords: Xiashi surgical
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Qinzhuliangxue Keli (Experimental): Qinzhuliangxue Keli(common name: QZLX particles, shenzhen China resources san-jiu pharmaceutical trading co., LTD.), loratadine tablets placebo (common name: LLTD piece, Shanghai schering pharmaceutical co., LTD.)
  Interventions: Drug: Furoic acid loperamide hydrochloride cream; Drug: Mullite ointment; Drug: 3% boric acid solution; Drug: Zine oxide
- loratadine tablets (Active Comparator): Qinzhuliangxue Keli placebo (common name: QZLX particles, shenzhen China resources san-jiu pharmaceutical trading co., LTD.),Loratadine tablets (common name: LLTD piece, Shanghai schering pharmaceutical co., LTD.).
  Interventions: Drug: Furoic acid loperamide hydrochloride cream; Drug: Mullite ointment; Drug: 3% boric acid solution; Drug: Zine oxide
- Qinzhuliangxue and loratadine (Active Comparator): Qinzhuliangxue Keli (common name: QZLX particles, shenzhen China resources san-jiu pharmaceutical trading co., LTD.), loratadine tablets (common name: LLTD piece, Shanghai schering pharmaceutical co., LTD.).
  Interventions: Drug: Furoic acid loperamide hydrochloride cream; Drug: Mullite ointment; Drug: 3% boric acid solution; Drug: Zine oxide

INTERVENTIONS:
Drug: Furoic acid loperamide hydrochloride cream — Apply to lesion area without erosion, drainage, 1 times a day, continuous use 1 week after according to disease reduction or withdrawal, the longest do not exceed 4 weeks. Pure dry area or no skin itching area should not be applied.
Drug: Mullite ointment — Applies to a blister, pustule, erosion, ulcer, leaking or comorbid folliculitis, in skin lesions of 2 times a day, 5 days for one period of treatment, but for two consecutive period of treatment
Drug: 3% boric acid solution — 3% boric acid solution is suitable for the erosion seepage skin, can open intermittent shi fu, 5-10 min each time, 2 times daily or several times.
Drug: Zine oxide — In wet apply the break to zinc oxide preparation for external use only, when erosion seepage control is disabled in skin lesions.

SUMMARY:
On the basis of Xiashi skin surgery clinical experience, this project adopts the multicenter, randomized, double-blind, controlled trial of design type. Objective, normative evaluation of traditional Chinese medicine cool blood latent town effectiveness of therapeutic regimen in the treatment of eczema, security, and control of the relapse of situation, provide high-level evidence-based basis for traditional Chinese medicine treatment of eczema, aims to form suitable for popularization and application of traditional Chinese medicine in the treatment of eczema.

ELIGIBILITY:
Inclusion Criteria:

* accord with standard of syndrome differentiation of traditional Chinese medicine (blood hot sheng) and western medicine diagnostic criteria (subacute eczema);
* age between 18-65 years old, gender, ethnic unlimited;
* agreed to participate in clinical trials can observe and cooperate with the visitor on schedule;
* volunteered for this study and obtain informed consent will be;
* lesion area of about 5-30% of surface area (BSA) were (containing 3% and 3%, palm measurement method)
* IGA scale of 1 to 3 points (including);
* her lesions mainly located in the trunk and limbs (or);
* Women HCG negative;

Exclusion Criteria:

* known to the study of drug allergy to any of the components;
* previous or current with any may affect the results of systemic disease, or other activity of skin diseases (such as: psoriasis);
* has a liver and kidney function is not complete, liver damage of ALT and AST > 1.5 times the upper limit of normal, renal BUN > 1.5 times the upper limit of normal or creatinine > 1.5 times the upper limit of normal value;
* QTcB or QTcF acuity 450 milliseconds. For subjects QTc acuity bundle branch block 480 milliseconds.
* prior or current with clinical significance of cardiovascular, lung disease, gastrointestinal tract, liver, kidney, blood, nerve abnormalities or mental disease;
* breast-feeding or plan to pregnant women during test;
* skin area score > 30%;
* eosinophil count score > 10%
* for nearly two weeks taking corticosteroids or a week, both inside and outside with corticosteroid preparation;
* three months received study medication or other participated in other clinical subjects;
* for any reason cannot cooperate research, for example: how language understanding, not to research centers, etc.;
* Researchers believe can bring obvious risk patients or confuse the results of the study, which should rule out other conditions or disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Eczema Area and Severity Index (EASI) score | Baseline and up to week 4 of the follow up phase

SECONDARY OUTCOMES:
Dermatology life quality index (DLQI) | Baseline and up to week 4 of the follow up phase
Change in Itching degree score | Baseline and up to week 4 of the follow up phase